CLINICAL TRIAL: NCT04325737
Title: A Randomized, Double-blind, Placebo-controlled, Multiple Oral Dose Study Assessing the Safety and Tolerability of SEP-363856 in Japanese Subjects With Schizophrenia
Brief Title: Study Assessing the Safety, Tolerability, and Pharmacokinetics of SEP-363856 in Japanese Male and Female Subjects With Schizophrenia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sumitomo Pharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DA801102
Record Dates: First submitted 2020-03-23; First posted 2020-03-30 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — SEP-363856

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SEP-363856 (Experimental)
  Interventions: Drug: SEP-363856
- Placebo (Placebo Comparator): Placebo will be orally administered according to the same administration schedule as the SEP-363856 group in each cohort.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SEP-363856 — Dosing of the SEP-363856 group in Cohort 1 will be initiated at 50 mg SEP-363856 as an oral once daily dose for 3 consecutive days, followed by 75 mg SEP-363856 as an oral once daily dose for 4 consecutive days, and followed by 100 mg SEP-363856 as an oral once daily dose for 7 consecutive days. The SEP-363856 group in Cohort 2 will be dosed at 25 mg SEP-363856 as an oral once daily dose for 3 consecutive days, followed by 50 mg SEP-363856 as an oral once daily dose for 3 consecutive days, followed by 75 mg SEP-363856 as an oral once daily dose for 4 consecutive days, and followed by 100 mg SEP-363856 as an oral once daily dose for 7 consecutive days.
  Arms: SEP-363856
Drug: Placebo — Placebo will be orally administered according to the same administration schedule as the SEP-363856 group in each cohort.
  Arms: Placebo

SUMMARY:
This is a multiple oral dose, randomized, double-blind, placebo-controlled study assessing the safety, tolerability and pharmacokinetics (PK) of SEP-363856 when administered qhs to Japanese subjects with schizophrenia.

DETAILED DESCRIPTION:
This multicenter study will be conducted in 2 cohorts (Cohort 1 and 2). Cohort transition will be determined by the Safety Review Team (SRT) before the start of Cohort 2.

For each cohort, the target number of subjects completing the treatment period is defined as 8 for SEP-363856 group and 4 for placebo group. Subjects will be randomly assigned to either group. Dosing of the SEP-363856 group in Cohort 1 will be initiated at 50 mg SEP-363856 as an oral once daily dose for 3 consecutive days, followed by 75 mg SEP-363856 as an oral once daily dose for 4 consecutive days, and followed by 100 mg SEP-363856 as an oral once daily dose for 7 consecutive days. The SEP-363856 group in Cohort 2 will be dosed at 25 mg SEP-363856 as an oral once daily dose for 3 consecutive days, followed by 50 mg SEP-363856 as an oral once daily dose for 3 consecutive days, followed by 75 mg SEP-363856 as an oral once daily dose for 4 consecutive days, and followed by 100 mg SEP-363856 as an oral once daily dose for 7 consecutive days. In the placebo group, placebo will be orally administered according to the same administration schedule as the SEP-363856 group in each cohort.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who voluntarily provide written consent to participate in the study. If the subject is considered a minor at the time of collection of the informed consent, written consent will be obtained from a legally acceptable representative (guardian) in addition to that obtained from the subject.
2. Subject who has schizophrenia diagnosed by DSM-5, diagnostic criteria, and in the opinion of the Investigator has been clinically stable.
3. Subject who has body weight >= 40.0kg and body mass index (BMI) >= 18.5.
4. Female subjects who are premenopausal and of childbearing potential must have a negative serum pregnancy test result.
5. Female subjects who are of childbearing potential and male subjects whose partners are of childbearing potential must agree to use adequate and reliable contraception.

other

Exclusion Criteria:

1. Subjects who experienced an acute exacerbation of psychosis requiring change in antipsychotic medication (with reference to drug or dose) within 90 days before screening.
2. Subjects who become strongly affected by potent central nervous system depressants (including barbiturate) as considered by the Investigator.
3. Subjects who have any clinically significant unstable medical condition or any clinically significant chronic disease that in the opinion of the Investigator, would limit the subject's ability to complete and/or participate in the study.
4. Subjects with active suicidal ideation or those with a suicide attempt history.
5. Subjects with a history or complication(s) of hypersensitivity to any medication.
6. Subjects with a history or complication(s) of malignant tumor within 5 years before screening, except for adequately treated basal cell or squamous cell skin cancer or in situ cervical cancer. Pituitary tumors of any duration are excluded.
7. Subjects who have previous or existing infection with human immunodeficiency virus (HIV) at screening.
8. Subjects who have a positive syphilis serological test, Hepatitis B virus surface (HBs) antigen or Hepatitis C virus (HCV) antibody at screening.

other

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2020-03-31 (Actual); Primary Completion 2020-08-07 (Actual); Study Completion 2020-08-07 (Actual)

PRIMARY OUTCOMES:
Frequency of AEs, serious adverse events (SAEs), and AEs resulting in study discontinuation | 18 days
  adverse events (AEs), serious adverse events (SAEs) in cohort 1.
Frequency of AEs, serious adverse events (SAEs), and AEs resulting in study discontinuation | 21 days
  adverse events (AEs), serious adverse events (SAEs) in cohort 2.

SECONDARY OUTCOMES:
Plasma concentrations of SEP-363856 and its metabolite SEP-363854 | 18 days
  Plasma concentrations in cohort 1.
Plasma concentrations of SEP-363856 and its metabolite SEP-363854 | 21 days
  Plasma concentrations in cohort 2.

CONTACTS AND LOCATIONS:
Locations (8):
- Japan (8):
  - Shiranui Hospital, Omuta-shi, Fukuoka
  - Nishiurakai Keihan Hospital, Osaka-Fu, Moriguchi-shi
  - Mental Support SOYOKAZE Hospital, Ueda-shi, Nagano
  - NHO Ryukyu Hospital, Kunigami-gun, Okinawa
  - NHO Hizen Psychiatric Center, Kanzaki, Saga-ken
  - Rainbow & Sea Hospital, Karatsu-shi, Saga-ken
  - Inuo Mental Care Hospital, Tosu, Saga-ken
  - Kuramitsu Hospital, Fukuoka

IPD SHARING:
Plan to Share IPD: Undecided